CLINICAL TRIAL: NCT04004260
Title: Cognitive Behavior Therapy Based Self-help Delivered Via the Internet for Tinnitus Sufferers: Efficacy Trial in the U.S. Population
Brief Title: CBT-based Internet Intervention for Adults With Tinnitus in the United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lamar University (Other)
Responsible Party: Principal Investigator, Vinaya Manchaiah, Jo Mayo Endowed Professor, Lamar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21DC017214 (NIH)
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: The experimental group will initially undergo the ICBT intervention while the control group are monitored weekly. Once the experimental group has completed the intervention, the control group will undertake the ICBT intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention offered is a guided Internet-based CBT intervention. The intervention is similar to a self-help program, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is a 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice the techniques learned.
  Interventions: Behavioral: Internet-based Cognitive Behavior Therapy
- Weekly check-in control group (Other): The weekly check-in control group will be monitored weekly by means of the Tinnitus Handicap Inventory-Screening version (THI-S) and the Tinnitus Qualities Questionnaire (TQQ). Once the experimental group completes the ICBT intervention, the control group undertake the same ICBT intervention.
  Interventions: Behavioral: Internet-based Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavior Therapy — The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.
  Other Names: ICBT

SUMMARY:
Nearly 50 million people in the U.S. experience tinnitus, of which about 20 million people have burdensome chronic tinnitus. Tinnitus can be very debilitating as many aspects of daily life can be affected, such as sleep, mood, and concentration. Currently, there is no cure for tinnitus. Pharmacological or sound-therapy based interventions are sometimes provided, but may be of limited value to certain individuals. Research suggests that Cognitive Behavior Therapy (CBT) based approaches have the most evidence of effectiveness in the management of tinnitus. However, CBT is rarely offered in the U.S. (less than 1%), partly attributed to a lack of trained professionals who can deliver CBT. To improve access to CBT for tinnitus, and online CBT program has been developed. The purpose of this study is to determine the feasibility and efficacy of a CBT Internet-based intervention for adults with tinnitus in the United States.

DETAILED DESCRIPTION:
Objective: This study aims to determine the feasibility and efficacy of an Internet-based Cognitive Behavior Therapy (ICBT) in reducing the impact associated with tinnitus in the United States.

Hypothesis: It is hypothesized that ICBT will result in reduced tinnitus-related distress, decreased sleep disturbance, decreased anxiety and depression, and improved health-related quality of life in a treatment group as compared with adults in the weekly check-in control-group in the U.S. population. The investigators also hypothesize that these results will be stable in both short- and long-term post-intervention.

Design: A two-armed Randomized Control Trial (RCT), with a one-year follow-up design will be used to evaluate the efficacy of ICBT on tinnitus distress.

Setting: This will be an Internet-based study for adults with tinnitus living in the State of Texas, USA.

Participants: Eligible participants will include adults with tinnitus for a minimum period of 3 months with internet access and no major medical or psychiatric conditions. 80 participants will be recruited for each group and will be randomly assigned using a computer-generated randomization schedule by an independent research assistant after being pre-stratified for language and tinnitus severity.

Intervention: The intervention offered is a guided CTB-based internet intervention (ICBT), providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.

Outcome measures: The main outcome measure is the Tinnitus Functional Index (TFI). Secondary outcome measures are the Tinnitus and Hearing Survey (THS), Tinnitus Cognition Questionnaire (TCQ), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), Insomnia Severity Index (ISI), and EuroQol EQ-5D-5L VAS.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years and older living in the State of Texas, USA;
2. the ability to read and type in English or Spanish;
3. no barriers to using a computer (e.g. no significant fine motor control or visual problems);
4. Internet and e-mail access and the ability to use it;
5. commitment to completing the program;
6. completion of the online screening and outcome questionnaires;
7. agreeing to participate in either group and be randomized to one of these groups;
8. understanding and working towards the end goal of reducing the impact and distress of tinnitus, although the strength of the tinnitus may remain the same;
9. be available for 12 months after starting the study to complete a 1-year follow-up questionnaire;
10. suffering with experiencing tinnitus for a minimum period of 3 months; and
11. tinnitus outcome measure scores indicating the need for tinnitus care [25 or above on the Tinnitus Functional Index (TFI)].

Exclusion Criteria:

1. reporting any major medical or psychiatric conditions;
2. reporting pulsatile, objective or unilateral tinnitus, which has not been investigated medically;
3. tinnitus as a consequence of a medical disorder, still under investigation; and
4. undergoing any other tinnitus therapy while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Manchaiah, PhD, Principal Investigator — Lamar University
Locations (1):
- Lamar University, Beaumont, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are openly available in Figshare at http://doi.org/10.6084/m9.figshare.13646012
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available now
Access Criteria: Data are openly available
URL: http://doi.org/10.6084/m9.figshare.13646012

REFERENCES:
- [Derived] W Beukes E, Andersson G, Fagelson M, Manchaiah V. Internet-Based Audiologist-Guided Cognitive Behavioral Therapy for Tinnitus: Randomized Controlled Trial. J Med Internet Res. 2022 Feb 14;24(2):e27584. doi: 10.2196/27584. PMID 35156936
- [Derived] Beukes EW, Andersson G, Manchaiah V. Patient Uptake, Experiences, and Process Evaluation of a Randomized Controlled Trial of Internet-Based Cognitive Behavioral Therapy for Tinnitus in the United States. Front Med (Lausanne). 2021 Nov 17;8:771646. doi: 10.3389/fmed.2021.771646. eCollection 2021. PMID 34869490
- See also: Related Info — http://www.tacklingtinnitus.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 315 participants completed the informed consent and completed the pre-intervention screening measures. However, 157 participants were excluded (49 participants reported high depression and/or positive answers to self-harm questions, 37 participants had low tinnitus severity, 71 participants resided outside the state/country) and the remaining 158 were included in the study.
Period: Overall Study
Arm/Group | Experimental Group | Weekly check-in Control Group
Started | 79 | 79
Completed | 37 | 47
Not Completed | 42 | 32
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Lost to Follow-up | 22 | 12
Not completed — Did not engage in intervention | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Weekly check-in Control Group | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (13) | 58 (11) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 40 | 38 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 70 | 68 | 138
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 2 | 4
  White | 74 | 74 | 148
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 79 | 79 | 158
Tinnitus Functional Index (TFI) [Mean (Standard Deviation); unit: score on a scale] | 54.04 (17.85) | 53.93 (17.32) | 53.98 (17.53)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index (TFI) - Measure of Tinnitus Distress
Description: The Tinnitus Functional Index (TFI) is a 25-item questionnaire that evaluates tinnitus distress. The total possible score ranges from 0-to-100 with higher scores indicate more severe tinnitus distress (i.e., worse outcome). Scores >25 indicate tinnitus is a significant problem requiring tinnitus intervention.
Time Frame: T0: Baseline, T1: Post-intervention after the experimental group completed the intervention, T2: Post-intervention after control group completed intervention; T3: 2-months post-intervention
Population: 79 participants started the trial in both the experimental group and control group 41 participants from the experimental group and 66 from the control group completed the post-intervention measure at T137 participants from the experimental group and 47 from the control group completed the post-intervention measure at T2 37 participants from the experimental group and 25 from the control group completed the 2-month post-intervention measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 54.04 (17.85) | 53.93 (17.32)
  T1: Post-intervention for experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for experimental group | 29.44 (19.60) | 47.35 (21.25)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 25.10 (19.46) | 38.50 (21.36)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 25.10 (19.46) | 32.82 (14.70)

2. Secondary Outcome: Tinnitus Cognition Questionnaire (TCQ); Measure of Tinnitus Cognition
Description: Tinnitus Cognition Questionnaire (TCQ) is a 26-item questionnaire that assesses positive and negative cognitions associated with tinnitus. The first 13 items refer to negative thoughts and the second 13 items refer to positive thoughts. Responses are marked on a five-point Likert scale (0 to 4). The negative items (1-13) are scored 0-4, whereas the positive items (14-26) are reverse-scored: 4-0. The scoring procedure involves the simple addition of the number circled by the respondent for items 1-13 and the addition of reverse-scored items 14-26. The total score of the TCQ has a potential range from 0 to 104. A high score represents a greater tendency to engage in negative cognitions (i.e., worse outcome) in response to tinnitus and low engagement in positive cognitions.
Time Frame: Baseline, Post-intervention (8-weeks from baseline), 2-months post-intervention (16 weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 39.63 (17.38) | 37.95 (14.54)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 26.03 (15.58) | 26.03 (16.80)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 40.57 (15.72) | 32.26 (15.54)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 40.57 (15.72) | 28.55 (17)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-9); Measure of Depression
Description: Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that assesses depression severity. Responses are marked on a four-point Likert scale (0 to 3). The total score can range from 0 to 27 with higher scores indicating more severe depression (i.e., worse outcome).
Time Frame: Baseline, Post-intervention (8-weeks from baseline), 2-months post-intervention (16 weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 5.54 (4.17) | 5.42 (4.1)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 4.41 (4.74) | 5.91 (4.35)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 3.17 (4.01) | 4.20 (3.8)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 3.17 (4.01) | 3.70 (4.73)

4. Secondary Outcome: Generalized Anxiety Disorder (GAD-7); Measure of Anxiety
Description: Generalized Anxiety Disorder (GAD-7) is a 7-item questionnaire that assesses the severity of anxiety. Responses are marked on a four-point Likert scale (0 to 3). The total score can range from 0 to 21 with higher scores indicating more severe anxiety (i.e., worse outcome).
Time Frame: Baseline, Post-intervention (8-weeks from baseline), 2-months post-intervention (16 weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 5.97 (4.22) | 5.23 (4.29)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 4.8 (4.84) | 5.35 (4.59)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 3.77 (4.65) | 3.77 (3.52)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 3.77 (4.65) | 5.17 (5.58)

5. Secondary Outcome: Insomnia Severity Index (ISI); Measure of Insomnia
Description: Insomnia Severity Index (ISI) is a 7-item questionnaire that evaluates the severity of insomnia. Responses are marked on a five-point Likert scale (0 to 4). The total score can range from 0 to 28 with higher scores indicating more severe insomnia (i.e., worse outcome).
Time Frame: Baseline, Post-intervention (8-weeks from baseline), 2-months post-intervention (16 weeks from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 10.18 (5.99) | 9.92 (5.71)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 5.98 (4.8) | 9.97 (6.39)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 4.97 (5.0) | 7.70 (5.56)
  T3: 2-months post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-months post-intervention | 4.97 (5.0) | 5.77 (6.24)

6. Secondary Outcome: EuroQol EQ-5D-5L VAS Scores; Measure of Health-related Quality of Life
Description: EQ-5D-5L VAS is a single questionnaire that evaluates the health-related quality of life. Responses are marked on a 0-100 scale with higher scores indicate the higher overall health-related quality of life (i.e., better outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 78.23 (13.14) | 75.51 (13.96)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 79.68 (15.66) | 76.02 (13.7)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 80.79 (16.16) | 78.52 (13.29)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 80.79 (16.16) | 78.05 (21.44)

7. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Tinnitus Sub-scale; Measure of Tinnitus Problem
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problems and the ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 16 with higher scores indicating more tinnitus problem (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 5.80 (3.9) | 5.51 (3.52)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 2.68 (2.47) | 5.31 (3.82)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 2.35 (3.4) | 3.46 (3.10)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 2.35 (3.4) | 2.86 (3.68)

8. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Hearing Sub-scale; Measure of Hearing Problem
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problems and the ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). However, the scores for this specific sub-scale can range from 0 to 16 with higher scores indicating more hearing problem (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | 6.89 (4.5) | 7.30 (4.79)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | 3.83 (3.65) | 7.29 (4.94)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | 3.21 (3.2) | 6.46 (4.05)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | 3.21 (3.2) | 4.14 (3.37)

9. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Sound Tolerance Sub-scale; Measure of Sound Tolerance
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problems and the ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). However, the scores for this specific sub-scale can range from 0 to 8 with higher scores indicating more sound tolerance problem (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Control Group
Number analyzed (Participants) | 79 | 79
score on a scale
  T0: Baseline | .87 (1.3) | .8 (1.1)
  T1: Post-intervention for the experimental group: number analyzed (Participants) | 41 | 66
  T1: Post-intervention for the experimental group | .54 (.84) | 1.0 (1.3)
  T2: Post-intervention for the control group: number analyzed (Participants) | 37 | 47
  T2: Post-intervention for the control group | .47 (.79) | .76 (1.14)
  T3: 2-month post-intervention: number analyzed (Participants) | 37 | 25
  T3: 2-month post-intervention | .47 (.79) | .64 (.9)

ADVERSE EVENTS:
Time Frame: T0: Baseline, T1: Post-intervention after the experimental group completed the intervention, T2: Post-intervention after control group completed intervention; T3: 2-months post-intervention
Description: Our definition of adverse events is the same as clinical trials.gov.
Arm/Group | Experimental Group | Weekly check-in Control Group
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79

LIMITATIONS AND CAVEATS:
The study was done during the height of the COVID-19 pandemic, during a time where day-to-day living was disrupted for most people. This may have been one of the key reasons for poor engagement with the intervention and poor compliance with the completion of outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT04004260/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT04004260/ICF_001.pdf